CLINICAL TRIAL: NCT00465972
Title: A Randomized, Double-blind, Placebo Controlled Study to Assess the Efficacy and Safety of Doxepin and Temazepam in HIV Seropositive Patients With Insomnia.
Brief Title: The Treatment of Insomnia in Patients With HIV Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8899
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-05

CONDITIONS: HIV Infections; Insomnia
Keywords: HIV; Insomnia; Cytokines; Adherence
MeSH Terms: conditions — HIV Infections; Sleep Initiation and Maintenance Disorders | interventions — Doxepin; Temazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Active Comparator): Doxepin
  Interventions: Drug: Doxepin
- 3 (Active Comparator): Temazepam
  Interventions: Drug: Temazepam

INTERVENTIONS:
Drug: Doxepin — Doxepin 10 mg po nightly x duration of study length OR Temazepam 15 mg po nightly x duration of study length OR Placebo nightly x duration of study length
  Arms: 2
Drug: Temazepam — Temazepam capsule 15 mg po nightly x duration of study
  Arms: 3
Drug: Placebo — Placebo capsule nightly for duration of study
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the efficacy of two commonly prescribed sleep aids for use in patients who are HIV positive and suffer from insomnia.

DETAILED DESCRIPTION:
Insomnia is a disorder defined as persistent difficulty falling asleep, staying asleep or non-restorative sleep which is associated with diminished daytime function without any identifiable underlying cause. This condition is extremely common among HIV infected individuals and can lead to significant distress and reduction in the quality of life. The mechanisms for disrupted sleep in this population are diverse, including potential direct effects of the tat protein upon the sleep centers in the central nervous system. Insomnia has been documented to be one of the most common psychiatric disorders in HIV disease, but no trial has systematically examined the efficacy of available hypnotic agents, which are commonly used in this population.

Comparison(s): Two commonly prescribed hypnotic agents used for insomnia will be compared to placebo over a 6 month treatment study.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia
* HIV Seropositive
* Stable HIV Disease

Exclusion Criteria:

* Other psychiatric illnesses
* Unstable HIV disease

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Krystal, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Reid S, Dwyer J. Insomnia in HIV infection: a systematic review of prevalence, correlates, and management. Psychosom Med. 2005 Mar-Apr;67(2):260-9. doi: 10.1097/01.psy.0000151771.46127.df. PMID 15784792
- [Derived] Low Y, Preud'homme X, Goforth HW, Omonuwa T, Krystal AD. The association of fatigue with depression and insomnia in HIV-seropositive patients: a pilot study. Sleep. 2011 Dec 1;34(12):1723-6. doi: 10.5665/sleep.1446. PMID 22131611

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from an HIV clinic in the Department of Internal Medicine, Duke University Medical Center
Pre-assignment Details: We initially planned to have 3 arms: placebo, temazepam, and doxepin. However, based on the rate of recruitment, we limited the study to 2 arms: placebo and temazepam.
  Screening was carried out which included medical, and psychiatric, and sleep assessments.
Groups:
- Placebo: One sugar pill taken orally at bedtime for duration of the participant's involvement.
- Temazepam: One 15 mg temazepam pill taken orally at bedtime for the duration of the participant's involvement.
Period: Overall Study
Arm/Group | Placebo | Temazepam
Started | 20 | 24
Completed | 18 | 23
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: 1 sugar pill taken nightly at bedtime.
- Temazepam: 1 15 mg pill taken nightly at bedtime.
- Total: Total of all reporting groups
Arm/Group | Placebo | Temazepam | Total
Number analyzed (Participants) | 18 | 23 | 41
Age Continuous [Mean (Standard Deviation); unit: Years] | 48.46 (5.1) | 47.8 (7.9) | 48.1 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 10 | 13 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 22 | 38
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Insomnia Severity Index [Mean (Standard Deviation); unit: Scores on a scale] — Measures the severity of insomnia on 7 items, with a rating of 0 (low severity) to 4 (high severity). Total range for the index is 0-28; with 28 being the most severe.
  Scores on a scale | 17.7 (4.9) | 16.6 (5.1) | 17.1 (5.0)
Piper Fatigue Scale [Mean (Standard Deviation); unit: Scores on a scale] — A 22 item survey measuring level of fatigue. Subjects answer each item on a scale of 1 - 10, with 1 being low fatigue, and 10 being severe fatigue. Total range of overall score is 22-220, with 220 being severe fatigue.
  Scores on a scale | 138 (42) | 114 (48) | 116 (45)

OUTCOME MEASURES:

1. Primary Outcome: Response: Change in Insomnia Severity Rating Scale at 3 Months.
Description: Insomnia Severity Index; It is a measure of Insomnia Severity; A higher number indicates greater severity of insomnia. Range of possible score totals is 0-28.
Time Frame: Baseline and 3 months
Population: This is the LOCF population
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: 1 sugar pill taken orally at bedtime.
- Temazepam: 1 15 mg pill of temazepam taken orally at bedtime.
Arm/Group | Placebo | Temazepam
Number analyzed (Participants) | 18 | 23
units on a scale | 0.72 (6.1) | -4.01 (5.3)

2. Secondary Outcome: Change in Piper Fatigue Scale at 3 Months
Description: A 22 item scale measuring level of fatigue, with possible totals ranging from 22-220. A higher number indicates greater severity of fatigue.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: 1 sugar taken nightly at bedtime.
Arm/Group | Placebo | Temazepam
Number analyzed (Participants) | 18 | 23
units on a scale | 12 (6.1) | 17 (5.3)

ADVERSE EVENTS:
Groups:
- Temazepam: 1 15 mg pill taken orally, nightly, at bedtime.
Arm/Group | Placebo | Temazepam
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/23
Other Adverse Events (participants affected / at risk) | 2/18 | 4/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | Temazepam (N=23)
dry mouth (Nervous system disorders) | 1 (1) | 3 (3)
sedation (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No